CLINICAL TRIAL: NCT05232201
Title: Elucidation of Vitamin D Levels and Heart Rate Variability Influence on Endothelial Function Via Renin Angiotensin Aldosterone System Augmentation in Obstructive Sleep Apnea
Brief Title: Vitamin D Levels and Heart Rate Variability on Endothelial Function Via RAAS Augmentation in OSA
Acronym: RAAS_OSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Sponsor
Other Study IDs: RAAS in OSA
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of obstructive sleep apnea (OSA) in contributing to hyperaldosteronism, which can lead to increased morbidity and mortality, is less well-established. The vitamin D levels and sympathetic activity of patients with obesity and OSA have not been explored in detail. In this cohort, the role of vitamin D and sympathetic activity, either individually or in combination, on augmenting the renin-angiotensin-aldosterone system (RAAS) causing more endothelial dysfunction remains elusive.

We aim to evaluate renin angiotensin aldosterone system in OSA population; elucidate relationship between aldosterone and vitamin D levels in patients with OSA; and to determine association between aldosterone level and vitamin D deficiency with cardio-metabolic derangement in patients with OSA.

This is a cross-sectional study involving 150 patients confirmed to have OSA. Participants who fulfil study criteria and consent to study will have blood withdrawn for aldosterone, renin, 25OHD levels with bone profile, and metabolic profile; undergo ultrasound flow mediated dilatation of brachial artery to assess endothelial function; ultrasound of hepatobiliary system to assess fatty liver; 24-hour Holter monitoring to assess sympathetic function; WHOQOLBREF to assess quality of life and Pittsburgh Sleep Quality Index to assess sleep quality.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), which is closely related to obesity, is a chronic, serious and potentially life-threatening sleep-related breathing disorder, characterized by periodic narrowing and obstruction of the pharyngeal airway during sleep, occurring in 25% to 58% of men and 10% to 37% of women.

Untreated OSA leads to lost productivity and workplace accidents resulting in injury and fatality. Patients with OSA are involved in automobile accidents more frequently than other licensed drivers. OSA is also associated with long-term health complications, including metabolic disorders and cardiovascular diseases, which is the leading cause of death worldwide.

For decades, we have believed that the activation of RAAS, mainly in response to intravascular volume contraction, regulated the biosynthesis of aldosterone. There is growing evidence that suggests aldosterone secretion to be beyond RAAS regulation. There is new evidence that both plasma and urinary aldosterone concentrations are increased in people with obesity. This relationship, on the other hand, is less studied for patients with OSA, with equivocal data. Aldosterone levels contributed to severity of OSA in patients with primary aldosteronism and resistant hypertension. In a limited number of studies, primary aldosteronism was found to be more frequent in patients with OSA whereas patients with OSA had higher aldosterone levels and prevalence of PA.

Vitamin D plays an important role in calcium homeostasis and metabolism. It is involved in maintenance of calcium and phosphorus levels in the blood, and bone content. Vitamin D is also implicated in several non-skeletal conditions, such as cardiovascular disease, cancer, autoimmune disorders and diabetes mellitus. Vitamin D deficiency has been associated with worse cardiovascular outcomes. Vitamin D deficiency augments the RAAS leading to elevated aldosterone and lowered renin. This is supported by a reduction in aldosterone and an increase in plasma renin in patients with heart failure, arterial hypertension and primary aldosteronism when repleted with vitamin D.

Sympathetic and parasympathetic nervous system interactively regulate visceral functions to maintain the body homeostatic milieu, and to enable reaction and adaptation to external and internal stressor stimuli. Patients with OSA exhibit high levels of sympathetic activity during sleep as well as when awake. Aldosterone is found to augment sympathetic activity in patients with resistant hypertension.

Heart rate variability (HRV) is a method that involves analysis of different parameters based on time variation between successive heart beats. HRV reflects the relationship between sympathetic and parasympathetic nervous system, which is a good predictor of future cardiovascular problems.

Endothelial dysfunction is a known risk factor for cardiovascular events. Vitamin D is known to have vaso-protective effect, while vitamin D deficiency leads to endothelial dysfunction. Besides, vitamin D has an anti-inflammatory property and acts by suppressing pro-inflammatory markers to prevent endothelial dysfunction. Vitamin D also elicits anti-oxidant effects through upregulating expression of anti-oxidative enzymes.

We postulate that

1. patients with OSA have higher aldosterone levels compared to healthy population;
2. hyperaldosteronism is associated with more vitamin D deficiency in patients with OSA;
3. hyperaldosteronism and vitamin D deficiency are associated with more cardio-metabolic derangement in the OSA population.

Research objectives

1. To evaluate renin angiotensin aldosterone system in OSA population;
2. To elucidate relationship between aldosterone and vitamin D levels in patients with OSA;
3. To determine association between aldosterone level and vitamin D deficiency with cardio-metabolic derangement in patients with OSA

Methodology Patients who are more than 18 years of age from the community, hospitals and clinics in Kuching, Samarahan and Serian will be invited to participate in this part of study if they fulfil the study criteria, after informed consent. Sleep study results will be interpreted by respiratory physicians. The community will be reached out via research advertisement or poster on UNIMAS facebook page, or via community health screening.

Study participants will be approached by researchers to be recruited into the study. Informed consent will be obtained by principal investigator in research clinic of UNIMAS main campus or Sarawak General Hospital Endocrine clinic depending on the convenience of the study participants.

Study participants will be given sufficient time to consider their participation in the study. The expected duration of participation for each study participant is 2 days. STOP-BANG score and Epsworth Sleepiness Scale will be documented at baseline. Their socio-demographic data will be collected and anthropometric measurements documented. If the participant has underlying hypertension, duration of hypertension and type of anti-hypertensive medications will be recorded. Anti-hypertensive will be switched to those with least effect on aldosterone and renin for at least 2 weeks before the start of research. Seated clinic blood pressure will be measured using appropriately-sized cuff at each clinic visit after 5 minutes of rest. The mean of 2 readings will be recorded.

Approximately 20ml of blood will be taken for aldosterone, renin, 25(OH)D, calcium, albumin, phosphate, intact parathyroid hormone, renal profile, HbA1c, plasma glucose, lipid profile, and hsCRP. No blood specimens will be stored for future research.

Study participants will also fill in the World Health Organization abbreviated version of quality of life (WHOQOL-BREF) questionnaire to assess their quality of life with OSA, and Pittsburgh Sleep Quality Index (PSQI) to assess sleep quality.

All study participants will also undergo ultrasound flow-mediated dilatation of brachial artery to assess endothelial function. At the same setting, hepatobiliary ultrasound will be performed to detect presence of hepatic steatosis. This procedure will be performed and results analysed by radiologist.

All study participants will have Holter monitor attached for 24 hours to assess heart rate variability as indicator for SNS activity. HRV will be analyzed using time-domain analysis as indicator of SNS activity. The results will be analysed by cardiologist.

Risks Blood taking may produce discomfort, minor bleeding, small possibility of bruising and slight risk of infection at the site of venepuncture. Although rare, some may experience vasovagal symptoms with blood draw. Blood taking will be performed by trained medical personnel to minimize these risks. If bruising occurs, it will be treated with warm compress and this will resolve after a few days. In the rare occasion that an infection occurs at venepuncture site, it will be treated with antibiotics.

Benefits Through this study, study participants will be able to obtain information about their serum aldosterone, renin, bone parameters, metabolic markers, any presence of sleep apnea, metabolic-associated fatty liver disease and other cardio-metabolic indices for free. Researchers will be able to understand further the relationship between OSA and aldosterone regulation, as well as role of aldosterone in contributing to sympathetic nerve function, endothelial function and vitamin D levels among patients with OSA.

Study withdrawal Participants will be withdrawn if i) they do not come for every study visit, ii) they choose to withdraw their consent at any time, iii) the investigator deems that it is unsuitable for the participants to continue. All withdrawn participants will continue the routine care for their underlying disease conditions. Withdrawn participants will be replaced until sample size is adequate within the time frame. The study will be terminated or suspended if there are unanticipated problems involving risks to the study participants.

Confidentiality All information obtained in the study will be kept and handled in a confidential manner. All study participants will only be identified by patient ID made known only to the researchers. Blood samples collected will be labelled only with the patient ID. Study data will be stored in a locked cabinet of research clinic in UNIMAS main campus. Collected data will be kept for 7 years, after which will be shredded and destroyed. Study participants are given access to their personal information and study data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above
2. Obese (BMI>27.5kg/m2)
3. Confirmed OSA (AHI>5)

Exclusion Criteria:

1. Secondary causes of obesity, such as Cushing's syndrome or thyroid dysfunction
2. Secondary hypertension, including undergone treatment for primary aldosteronism
3. Chronic kidney disease (eGFR<30ml/min/1.73m2)
4. Recent myocardial infarct or stroke within 6 weeks prior to study
5. Congestive heart failure
6. Long-standing atrial fibrillation >12 months
7. On current CPAP use
8. On vitamin D supplements
9. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea confirmed on sleep study (AHI>5)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Renin angiotensin aldosterone system | 30 months
  To evaluate renin angiotensin aldosterone system in OSA population
Aldosterone and vitamin D levels | 30 months
  To elucidate relationship between aldosterone and vitamin D levels in patients with OSA
Aldosterone level and vitamin D deficiency with cardio-metabolic derangement | 30 months
  To determine association between aldosterone level and vitamin D deficiency with cardio-metabolic derangement in patients with OSA

CONTACTS AND LOCATIONS:
Overall Officials: Huai Heng Loh, Principal Investigator — Universiti Malaysia Sarawak
Locations (1):
- Universiti Malaysia Sarawak, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No